CLINICAL TRIAL: NCT00382642
Title: Pharmacological Treatment for Alcoholism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bankole Johnson (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Bankole Johnson, Chair of Psychiatry and NB Sciences, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AA010522-11 (NIH); R01AA010522 (NIH)
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Alcohol Dependence
Keywords: alcoholism, alcohol disorder, drinking,alcohol
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron; Cognitive Behavioral Therapy; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ondansetron (Experimental): Arm 1 = Ondansetron 4 mcg/kg b.i.d.+ Cognitive behavioral therapy
  Interventions: Drug: Ondansetron + Cognitive Behavioral Therapy
- Placebo (Placebo Comparator): Arm 2 = Placebo + Cognitive behavioral therapy
  Interventions: Drug: Placebo + Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Ondansetron + Cognitive Behavioral Therapy — 13 week outpatient trial
  Other Names: Zofran
  Arms: Ondansetron
Drug: Placebo + Cognitive Behavioral Therapy — 13 week outpatient trial
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn whether ondansetron is safe and effective in the treatment of alcohol dependence. We also want to learn whether the study drug ondansetron combined with Cognitive Behavioral Therapy will assist researchers to determine whether having a certain gene is responsible for determining how a person benefits or does not benefit from the use of ondansetron for alcohol dependence.

DETAILED DESCRIPTION:
This is a 13 week outpatient clinical trial. Participants will either receive ondansetron or placebo and behavioral therapy. There is a 1, 2, and 3 month post-study follow up visit.Screening for this study is initially done over the telephone and takes 15-20 minutes. If participants are eligible after the initial screen, they will be invited to come in for a more thorough in house screen which takes about 5 to 6 hours. The screening will include a physical exam, review of medical, alcohol and drug histories and blood collection. If participants are found to be eligible after the in house screen, they will be enrolled in the 13 week outpatient clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who have given written informed consent.
* Ages 18 years and above and, must weigh at least 40 Kg and no more than 140 Kg
* Good physical health as determined by a complete physical examination, an EKG within normal limits, and laboratory screening tests within acceptable parameters.
* Audit score equal or more than 8
* Current DSM-IV diagnosis of alcohol dependence
* Currently drinking equal or more than 14 alcohol units/week for women and equal or more than 21 alcohol units/week for men in the last 30 days.
* Provide evidence of stable residence in the last month prior to enrollment in the study, and have no plans to move in the next three months.
* The pregnancy test for females at intake must be negative. Additionally, women of childbearing potential must be using an acceptable form of contraception. These include: oral contraceptives, hormonal (levonorgestrel) or surgical implants, or barrier plus spermicide.
* Literate in English and able to read, understand, and complete the ratings scales and questionnaires accurately, follow instructions, and make use of the behavioral treatments.
* Answer an advertisement in the newspaper/radio/television, and express a wish to stop drinking.
* Willingness to participate in behavioral treatments for alcoholism.

Exclusion Criteria:

* Subjects who are legally mandated to participate in an alcohol treatment program.
* Any current axis I DSM IV psychiatric disorder other than alcohol or nicotine dependence
* Elevation of liver enzymes - (SGOT), serum glutamic pyruvic transaminase (SGPT), blood urea nitrogen (BUN), or lactate dehydrogenase (LDH) greater than four times the normal range, or clinically significant elevated direct bilirubin as deemed by the principal investigator.
* Severe alcohol withdrawal symptoms which in the physicians opinion requires inpatient treatment.
* Serious medical co-morbidity requiring medical intervention or close supervision, or any condition, which can interfere with the receipt of ondansetron.
* Severe or life-threatening adverse reactions to ondansetron or similar medication either in the past or during this clinical trial.
* Female patients who are pregnant, lactating, or not adhering to an acceptable form of contraception at any time during the study.
* Received inpatient or outpatient treatment for alcohol dependence within the last 30 days (support groups such as AA are not exclusionary).
* Compelled to participate in an alcohol treatment program to maintain their liberty.
* Members of the same household.
* Treated with any medications having a potential effect on alcohol consumption and related behaviors, or mood. These include: opiate antagonist (e.g. naltrexone), glutamate antagonists (e.g., acamprosate), serotonin re-uptake inhibitors (e.g. fluoxetine), serotonin antagonists (e.g. ritanserin or buspirone), other antidepressants (e.g. tricyclic antidepressants or monoamine oxidase inhibitors), dopamine antagonists (e.g. haloperidol), calcium channel antagonists (e.g. isradipine), or compounds with actions similar to disulfiram (antabuse) or nicotine.
* Before double-blind randomization, urine must be free of opiates, cocaine, amphetamines, barbiturates, benzodiazepines, prescription and non-prescription drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Self-reported measure of alcohol consumption (Drinks per Day, Drinks per Drinking Day, Percent Days Abstinent), CDT (ondansetron level), GGT, BAC | Throughout the study

SECONDARY OUTCOMES:
Pill count, CIWA-Ar, OCDS, Age of onset, SFQ, AASE, ADBS, CGI, TCI, MAC, attendace at psychosocial services | Throughout the study
  medication compliance, withdrawal, alcohol craving, social functioning and motivation

CONTACTS AND LOCATIONS:
Overall Officials: Bankole Johnson, M.D., Ph.D., Principal Investigator — University of Virginia
Locations (1):
- UVA Center for Addiction Research and Education, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Johnson BA, Seneviratne C, Wang XQ, Ait-Daoud N, Li MD. Determination of genotype combinations that can predict the outcome of the treatment of alcohol dependence using the 5-HT(3) antagonist ondansetron. Am J Psychiatry. 2013 Sep;170(9):1020-31. doi: 10.1176/appi.ajp.2013.12091163. PMID 23897038